CLINICAL TRIAL: NCT06782633
Title: Assessment of Deep Core Muscles, Postural Analysis, Functional and Mental Performance in Different Age Group of Asymptomatic Participants and Patients With Non-specific Low Back Pain
Brief Title: Deep Core Muscles and Biopsychosocial in Asymptomatic Adults and NSCLBP
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency); National Taiwan University (Other)
Responsible Party: Sponsor
Other Study IDs: 202012268RIND; MOST 111-2221-E-002-059 (Other Grant/Funding Number: National Science and Technology Council, Taiwan); MOST 112-2221-E-002-092 (Other Grant/Funding Number: National Science and Technology Council, Taiwan)
Record Dates: First submitted 2025-01-10; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Non-Spesific Chronic Low Back Pain; Aged

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non-specific chronic low back pain: Participants with non-specific chronic low back pain (CLBP) aged 20-65 years old were recruited from the community by posters. Non-specific chronic low back was defined as discomfort in the low back area, which persisted over a day during the past three months and was diagnosed as non-specific low back pain. Participants who 1) had gone through surgery at the low back or lower extremity; 2) presented neurological symptoms, such as numbness or tingling; 3) could not walk or stand independently; 4) had cancer; 5) had systemic inflammation, such as ankylosing spondylitis, rheumatoid arthritis, and systemic lupus erythematosus; 6) were in pregnancy were excluded from the study.
- Asymptomatic: Asymptomatic participants aged 20-65 years old were recruited from the community by posters. Participants who 1) had gone through surgery at the low back or lower extremity; 2) presented neurological symptoms, such as numbness or tingling; 3) could not walk or stand independently; 4) had cancer; 5) had systemic inflammation, such as ankylosing spondylitis, rheumatoid arthritis, and systemic lupus erythematosus; 6) were in pregnancy were excluded from the study.

SUMMARY:
The goal of this observational study is to (1) investigate age effects on core muscles, sensorimotor system, psychosocial factors in asymptomatic adults across years of age; (2) explore the differences in biopsychosocial factors between asymptomatic adults and people with non-specific chronic low back pain (NSCLBP); (3) study the correlations between biopsychosocial factors in people with NSCLBP.

The main questions it aims to answer :

1. Are the core muscles, lumbar propriocpetion, and psychological measures altered as age increases?
2. Do the core muscles, lumbar propriocpetion, functional performance, psychological measures, disability, and quality of life affected by NSCLBP?
3. following (2), if so, are there correlations between the measured biopsychosocial factors, disability, and quality of life in people with NSCLBP?

Researchers will compare between people with NSCLBP and age-matched asymptomatic participants across years of age to see if the effect of age and effect of NSCLBP existed in biopsychosocial factors.

Participants will

1. be observed by ultrasound image at the low back and abdominal areas to collect parameters related to trunk deep core muscles, such as changes in muscle thickness from resting state to contraction;
2. ungergo MRI examination to acquire image of deep core muscles;
3. perform lumbar repositioning test which quantifies the lumbar proprioception;
4. perform Timed Up-and-Go Test and Five-Times Sit-to-Stand test, which are used as a measurement of physically functional performance;
5. fill out the psychosocial questionnaires including: Patient-Reported Outcomes Measurement Information System Short Form Depression 4a and Anxiety 4a, Pittsburgh Sleep Quality Index, Pain Catastrophizing Scale, Fear-Avoidance Belief Questionnaire, Oswestry Disability Index, and Heath Survey Short Form-36.

ELIGIBILITY:
Inclusion Criteria:

* aged above 20 years old
* Non-specific chronic low back defined as discomfort in the low back area, which persisted over a day during the past three months and was diagnosed as non-specific low back pain.

Exclusion Criteria:

* history of surgery at the low back or lower extremity
* neurological symptoms, such as numbness or tingling
* not able to walk or stand independently
* cancer
* systemic inflammation, such as ankylosing spondylitis, rheumatoid arthritis, and systemic lupus erythematosus
* in pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Taiwanese people
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Deep core muscles thickness by USI | On the 1 day of data collection for all parameters.
  The deep core muscles, including transversus abdominis, psoas major, and multifidus, are observed by USI. During USI measurements, participants are instructed to perform specific movement within normal range of motion to activate muscles.
Deep core muscles thickness by MRI | On the 1 day of data collection for all parameters or the day arranged specifically for MRI.
  The deep core muscles, including transversus abdominis, psoas major, and multifidus, are observed by MRI. Data collected by MRI is analyzed through ImageJ.
Deep core muscles cross-sectional area | On the 1 day of data collection for all parameters or the day arranged specifically for MRI.
  The deep core muscles, including transversus abdominis, psoas major, and multifidus, are observed by MRI. Data collected by MRI is analyzed through ImageJ with threshold method, to acquire funcitonal cross-sectional area of core muscles.
Lumbar proprioception | On the 1 day of data collection for all parameters.
  Proprioception was evaluated by lumbar repositioning error with the Zebris motion analysis system (Zebris Medizintechnik GmbH, Isny, Germany). The smaller the error suggests the better proprioception. Repositioning test was performed in a standing position. Participants were first instructed and practiced anterior and posterior pelvic tilting with minimal paraspinal muscle activation, and the neutral position of the lumbar spine was identified. Then, anterior and posterior pelvis tilting to the half and maximal range were practiced with eyes closed. For the actual tests, participants performed 5 repetitions of half range of anterior tilt, back to neutral spine, half range of posterior tilt, and back to neutral spine position. The performance of the first repetition served as the reference for the repositioning test. The error between the reference and the following 4 repetitions indicated the proprioception of the lumbar spine.
Functional performance-Timed Up-and-Go | On the 1 day of data collection for all parameters.
  Timed-Up-and-Go (TUG) was adopted to test functional performance. A 10-foot walkway was set with a chair at one end and a mark on the other. Trunk muscle activation for stabilization, lower limb strength, and mobility were required to complete the test.
Functional performance-Five-Times Sit-to-Stnad | On the 1 day of data collection for all parameters.
  Five-Times Sit-To-Stand (5-STS) was adopted to test functional performance. Participants were asked to perform sit to stand for consecutive 5 repetitions as fast as possible. Trunk muscle activation for stabilization, lower limb strength, and mobility were required to complete 5-STS.
Psychological Distress | On the 1 day of data collection for all parameters.
  Psychological distress were evaluated with the Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form Depression 4a and Anxiety 4a, which included 4 questions for each domain. Raw scores of PROMIS Short Form Depression 4a and Anxiety 4a were transformed into T scores according to the scoring manual (HealthMeasures; HealthMeasures). Higher scores of PROMIS indicated a higher degree of depression or anxiety.
Sleep Quality | On the 1 day of data collection for all parameters.
  Sleep quality was examined with the Pittsburgh Sleep Quality Index (PSQI), a self-report questionnaire that assesses sleep quality over a 1-month time interval.
Cognition toward pain | On the 1 day of data collection for all parameters.
  Fear-Avoidance Beliefs Questionnaire (FABQ) and Pain Catastrophizing Scale (PCS) were filled out to quantify the cognition and behaviors toward pain. Higher scores on both questionnaires indicated greater fear or tendency to catastrophize.
Disability | On the 1 day of data collection for all parameters.
  Oswestry Disability Index (ODI) was used to measure the disability, which included 10 questions. The total scores of ODI ranged from 0 to 50 and higher scores indicated a higher extent of disability.
Quality of life | On the 1 day of data collection for all parameters.
  Short Form-36 (SF-36) questionnaire was used to assess physical, psychological, and social factors, whose dimensions include physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social function (SF), role emotional (RE), and mental health (MH). Standardized scores of each domain in SF-36 ranged from 0 to 100 and higher scores referred to higher satisfaction. Raw scores of each domain in SF-36 were standardized according to the SF-36 Health Survey Manual.

SECONDARY OUTCOMES:
VAS | On the 1 day of data collection for all parameters.
  Pain intensity is measured by Visual Analog Scale in which the 10 indicates the most severe pain participants can imagine.
Hip range of motion | On the 1 day of data collection for all parameters.
  Hip joint range of motion was measured, including extension, internal rotation, and external rotation.
Stability test | On the day of data collection for all parameters.
  Stability was examined by Shraman's test. There were five levels of movement tasks. Completing the tasks meanwhile maintaining spine stability was the required. The higher level completed indicates better stability.

CONTACTS AND LOCATIONS:
Locations (1):
- School and Graduate Institute of Physical Therapy, National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided